CLINICAL TRIAL: NCT03566238
Title: A Double-Blind, Randomized, Placebo-Controlled, Phase 3 Study to Demonstrate Efficacy and Safety of A4250 in Children With Progressive Familial Intrahepatic Cholestasis Types 1 and 2 (PEDFIC 1)
Brief Title: This Study Will Investigate the Efficacy and Safety of A4250 in Children With PFIC Types 1 or 2
Acronym: PEDFIC 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Albireo (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A4250-005
Record Dates: First submitted 2018-05-25; First posted 2018-06-25 (Actual); Results first posted 2021-09-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: PFIC1; PFIC2
Keywords: Pediatric; Cholestasis
MeSH Terms: conditions — Cholestasis | interventions — odevixibat

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Placebo-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A4250 low dose (Experimental): Capsules for oral administration (40 ug/kg) once daily for 24 weeks
  Interventions: Drug: A4250 (odevixibat)
- A4250 high dose (Experimental): Capsules for oral administration (120 ug/kg) once daily for 24 weeks
  Interventions: Drug: A4250 (odevixibat)
- Placebo (Placebo Comparator): Capsules for oral administration (to match active) once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: A4250 (odevixibat) — A4250 is a small molecule and selective inhibitor of ileal bile acid transporter (IBAT).
  Arms: A4250 high dose; A4250 low dose
Drug: Placebo — Placebo identical in appearance to active drug (A4250).
  Arms: Placebo

SUMMARY:
Double blind, randomized, placebo controlled, Phase 3 study to investigate the efficacy and safety of low doses and high doses of A4250 compared to placebo in children with progressive familial intrahepatic cholestasis (PFIC) types 1 and 2.

DETAILED DESCRIPTION:
Up to 50 sites in the following countries will take part in this study:

Australia, Belgium, Canada, France, Germany, Israel, Italy, Netherlands, Poland, Spain, Sweden, Turkey, United Kingdom, United States, and Saudi Arabia

ELIGIBILITY:
Key Inclusion Criteria:

* A male or female participant with a clinical diagnosis of PFIC Type 1 or 2 and with a body weight above 5 kg
* Participant must have clinical genetic confirmation of PFIC-1 or PFIC-2
* Participant must have elevated serum bile acid (s-BA) concentration
* Participant must have history of significant pruritus and a caregiver reported observed scratching in the eDiary
* Participant and/or legal guardian must sign informed consent (and assent) as appropriate.
* Participants will be expected to have a consistent caregiver(s) for the duration of the study
* Caregivers and age-appropriate participants (≥8 years of age) must be willing and able to use an eDiary device as required by the study

Key Exclusion Criteria:

* Participant with pathologic variations of the ABCB11 gene that predict complete absence of the bile salt export pump (BSEP) protein
* Participant with past medical history or ongoing presence of other types of liver disease including, but not limited to, the following:

  1. Biliary atresia of any kind
  2. Benign recurrent intrahepatic cholestasis, indicated by any history of normal s BAs
  3. Suspected or proven liver cancer or metastasis to the liver on imaging studies
  4. Histopathology on liver biopsy that is suggestive of alternate non-PFIC related etiology of cholestasis
* Participant with past medical history or ongoing chronic diarrhea
* Any participant with suspected or confirmed cancers except for basal cell carcinoma
* Participant with a past medical history of chronic kidney disease with an impaired renal function and a glomerular filtration rate <70 mL/min/1.73 m^2
* Participant with surgical history of disruption of the enterohepatic circulation (biliary diversion surgery) within 6 months prior to start of Screening Period
* Participant has had a liver transplant or a liver transplant is planned within 6 months of randomization
* Decompensated liver disease
* Participant suffers from uncontrolled, recalcitrant pruritic condition other than PFIC
* Participant who has been previously treated with an IBAT inhibitor whose pruritus has not responded to treatment

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Denver, Colorado
  - Emory University School of Medicine, Atlanta, Georgia
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center - Presbyterian Hospital Building, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine - Texas Children's Liver Center, Houston, Texas
- The Royal Children's Hospital, Melbourne, Australia
- Belgium (2):
  - UZ Leuven, Leuven
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- France (4):
  - University and Pediatric Hospital of Lyon, Bron
  - Universite Paris SUD - Hopitaux Universitaires Paris-Sud - Hopital Bicetre, Le Kremlin-Bicêtre
  - Hospital de la Timone, Marseille
  - Hospital Necker-Enfants maladies, Paris
- Germany (3):
  - Uniklinikum Essen- Kinderklinik II, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Kinderklinik Tübingen, Universitätsklinikum Tübingen, Tübingen
- Israel (3):
  - Rambam Medical Centre, Haifa
  - Shaare-Zedek Mc, Jerusalem
  - Schneider Children's Medical Center Of Israel, Petah Tikva
- Italy (3):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - University Hospital Of Padova, Padua
  - Ospedale Regina Margherita, Torino
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Universitair Medisch Centrum (UMC) Utrecht, Utrecht
- Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw, Poland
- King Faisal Specialist Hospital & Research Centre, Riyadh, Saudi Arabia
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
- Astrid Lindgren Children's Hospital, Karolinska University Hospital, Solna, Sweden
- Turkey (Türkiye) (5):
  - Gazi University, Ankara
  - Hacettepe University Faculty of Medicine, Ankara
  - Akdeniz University, Antalya
  - Istanbul University Medical Faculty, Istanbul
  - Inonu University Medical Faculty, Malatya
- United Kingdom (3):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Leeds General Infirmary, Leeds
  - Institute of Liver Studies - Kings College Hospital, London

REFERENCES:
- [Derived] Gwaltney C, Ivanescu C, Karlsson L, Warholic N, Kjems L, Horn P. Validation of the PRUCISION Instruments in Pediatric Patients with Progressive Familial Intrahepatic Cholestasis. Adv Ther. 2022 Nov;39(11):5105-5125. doi: 10.1007/s12325-022-02262-7. Epub 2022 Sep 6. PMID 36066745
- [Derived] Thompson RJ, Arnell H, Artan R, Baumann U, Calvo PL, Czubkowski P, Dalgic B, D'Antiga L, Durmaz O, Fischler B, Gonzales E, Grammatikopoulos T, Gupte G, Hardikar W, Houwen RHJ, Kamath BM, Karpen SJ, Kjems L, Lacaille F, Lachaux A, Lainka E, Mack CL, Mattsson JP, McKiernan P, Ozen H, Rajwal SR, Roquelaure B, Shagrani M, Shteyer E, Soufi N, Sturm E, Tessier ME, Verkade HJ, Horn P. Odevixibat treatment in progressive familial intrahepatic cholestasis: a randomised, placebo-controlled, phase 3 trial. Lancet Gastroenterol Hepatol. 2022 Sep;7(9):830-842. doi: 10.1016/S2468-1253(22)00093-0. Epub 2022 Jul 1. PMID 35780807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, double-blind, placebo-controlled study was conducted in children with progressive familial intrahepatic cholestasis (PFIC) at 33 study centers in 12 countries between 16 May 2018 and 28 July 2020.
Pre-assignment Details: The study included up to an 8-week screening period, a 24-week treatment period, and a 4-week follow-up period. A total of 62 participants were enrolled in the study.
Groups:
- A4250 Low Dose: Capsules for oral administration [40 microgram per kilogram (mcg/kg)] once daily for 24 weeks.
  A4250 (odevixibat): A4250 is a small molecule and selective inhibitor of ileal bile acid transporter (IBAT).
- A4250 High Dose: Capsules for oral administration (120 mcg/kg) once daily for 24 weeks.
  A4250 (odevixibat): A4250 is a small molecule and selective inhibitor of IBAT.
Period: Overall Study
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Started | 20 | 23 | 19
Received Treatment | 20 | 23 | 19
Completed | 15 | 18 | 16
Not Completed | 5 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 5 | 4 | 2
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all randomized participants who received at least 1 dose of study treatment.
Groups:
- A4250 Low Dose: Capsules for oral administration (40 mcg/kg) once daily for 24 weeks.
  A4250 (odevixibat): A4250 is a small molecule and selective inhibitor of IBAT.
- Total: Total of all reporting groups
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose | Total
Number analyzed (Participants) | 20 | 23 | 19 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 23 | 19 | 62
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.75 (3.853) | 3.86 (3.660) | 5.24 (4.188) | 4.25 (3.883)
Age, Customized [Count of Participants; unit: Participants]
  Age Category 1: 6 months to 5 years | 16 | 17 | 14 | 47
  Age Category 1: 6 to 12 years | 3 | 5 | 4 | 12
  Age Category 1: 13 to 18 years | 1 | 1 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 11 | 31
  Male | 12 | 11 | 8 | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 17 | 18 | 17 | 52
  Race: Black or African American | 0 | 2 | 0 | 2
  Race: Asian | 1 | 0 | 1 | 2
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Other | 2 | 3 | 1 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 1 | 0 | 0 | 1
  Ethnicity: Not Hispanic or Latino | 19 | 23 | 19 | 61
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 3 | 8
  United Kingdom | 5 | 6 | 2 | 13
  Saudi Arabia | 1 | 0 | 2 | 3
  Canada | 1 | 1 | 0 | 2
  Netherlands | 1 | 0 | 2 | 3
  Turkey | 1 | 7 | 3 | 11
  Poland | 2 | 0 | 1 | 3
  Italy | 1 | 1 | 0 | 2
  Israel | 1 | 0 | 1 | 2
  France | 1 | 3 | 1 | 5
  Australia | 1 | 0 | 0 | 1
  Germany | 2 | 3 | 4 | 9
Type of PFIC [Count of Participants; unit: Participants] — PFIC Type 1: Familial intrahepatic cholestasis-1 (FIC1) protein deficiency, PFIC Type 2: Bile salt export pump (BSEP) deficiency.
  Participants
    Type 1 | 5 | 7 | 5 | 17
    Type 2 | 15 | 16 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 70% Reduction in Fasting Serum Bile Acid (s-BA) Concentration From Baseline to the End of Treatment or Reaching a Level <=70 Micromoles Per Liter (Mcmol/L) After 24 Weeks of Treatment
Description: Fasting s-BA baseline was calculated as the average of the last 2 values prior to the first dose. The end value was the average of the values at Weeks 22 and 24 after the start of double-blind treatment. Participants who had at least 70% reduction in fasting s-BA from baseline to the end of treatment or reached <=70 mcmol/L after 24 weeks of treatment were considered as responder. Participants with missing average at the end of treatment were classified as non-responder. Percentages are rounded to hundredth decimal.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
percentage of participants | 0 [0.00 to 16.84] | 43.5 [23.19 to 65.51] | 21.1 [6.05 to 45.57]
Statistical Analysis 1: Comparison: Placebo vs A4250 Low Dose; Analysis was based on the Cochran Mantel Haenszel test adjusting PFIC type. A pooled analysis for the closed testing procedure was applied to control multiplicity. The 1-sided adjusted p-value for an individual dose was calculated as the maximum value of the unadjusted p-value for the pooled analysis and the unadjusted p-value for the individual doses. 1-sided adjusted p-value was reported; Test type: Superiority; p = 0.0015, Cochran-Mantel-Haenszel; percentage difference = 0.435, 95% CI 2-sided [0.2195 to 0.6551]
Statistical Analysis 2: Comparison: Placebo vs A4250 High Dose; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0174, Cochran-Mantel-Haenszel; percentage difference = 0.211, 95% CI 2-sided [0.021 to 0.4557]

2. Primary Outcome: Percentage of Positive Pruritus Assessments at the Participant Level Based on the Albireo Observer-Reported Outcome (ObsRO) Instrument Over the 24-Week Treatment Period
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least 1 point drop from baseline. The percentage of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant multiplied by 100.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Error); unit: percentage of assessments
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
percentage of assessments | 28.74 (5.209) | 58.31 (6.205) | 47.69 (8.110)
Statistical Analysis 1: Comparison: Placebo vs A4250 Low Dose; Analysis of the Proportion of Positive Pruritus Assessments at Participant Level over the 24-Week Treatment Period - Albireo ObsRO Instrument (AM and PM Scores); Test type: Superiority — Analysis of Covariance (ANCOVA) model including treatment, baseline pruritus score at AM and PM, PFIC type, and age category was used for treatment comparisons. A pooled analysis for the closed testing procedure was applied to control multiplicity. The 1-sided adjusted p-value for an individual dose was calculated as the maximum value of the unadjusted p-value for the pooled analysis and the unadjusted p-value for the individual doses. 1-sided adjusted p-value was reported; p = 0.0019, ANCOVA; Least Square (LS) mean difference = 28.23, 95% CI 2-sided [9.83 to 46.64], Standard Error of Mean 9.182
Statistical Analysis 2: Comparison: Placebo vs A4250 High Dose; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — An ANCOVA model including treatment, baseline pruritus score at AM and PM, PFIC type, and age category was used for treatment comparisons. A pooled analysis for the closed testing procedure was applied to control multiplicity. The 1-sided adjusted p-value for an individual dose was calculated as the maximum value of the unadjusted p-value for the pooled analysis and the unadjusted p-value for the individual doses. 1-sided adjusted p-value was reported; p = 0.0163, ANCOVA; LS mean difference = 21.71, 95% CI 2-sided [1.87 to 41.54], Standard Error of Mean 9.892

3. Secondary Outcome: Change From Baseline in Fasting Serum Bile Acid at Weeks 12 and 24
Description: Blood samples for analysis of s-BA were drawn at all visits. Participants were to fast (water intake only was permissible) for at least 4 hours prior to the collection of samples. Exceptions could be made for infants <12 months of age if they were unable to fast for the full 4 hours. Baseline was the average of the last 2 non-missing values of fasting s-BA concentration prior to the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment. Only participants with data collected at Baseline and Weeks 12 and 24 are reported.
Measure: Mean (Standard Error); unit: mcmol/L
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 17 | 20 | 16
mcmol/L
  Week 12 | 7.44 (24.588) | -113.70 (38.011) | -106.44 (41.201)
  Week 24: number analyzed (Participants) | 11 | 17 | 15
  Week 24 | 18.64 (31.559) | -145.03 (41.951) | -72.90 (52.617)

4. Secondary Outcome: Change From Baseline in Serum Alanine Aminotransferase (ALT) Concentration at Weeks 12 and 24
Description: Blood samples were collected to determine the ALT concentration. Baseline was the last available assessment before the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: units/L
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 18 | 22 | 18
units/L
  Week 12 | 1.7 (10.50) | -25.9 (23.36) | -13.8 (19.42)
  Week 24: number analyzed (Participants) | 11 | 17 | 15
  Week 24 | 3.7 (4.95) | -27.9 (17.97) | -25.3 (22.47)

5. Secondary Outcome: Change From Baseline in Growth Parameters at Weeks 12 and 24
Description: The change in the growth parameters was assessed using linear growth deficit [height (centimeter), weight (kilogram) and body mass index (BMI) (kg/meter square)] compared to standard growth curve (Z-score) calculated by using the software or methods from the centers for disease control (CDC) website for participants with age >=2 years old and from the world health organization website for participants with age <2 years old. Participants whose accurate age was not available, Z-score was not calculated. A Z-score indicated how many standard deviation's (SD) a participant's measurement (like height, weight and BMI), was from the average for their age and sex. A Z-score of 0 represents the median or 50th percentile, while positive or negative values show how far above or below average a measurement was. Baseline was the last available assessment before the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 18 | 22 | 16
z-score
  Height deficit: Week 12 | -0.03 (0.127) | 0.01 (0.108) | -0.06 (0.100)
  Height deficit: Week 24: number analyzed (Participants) | 12 | 17 | 15
  Height deficit: Week 24 | -0.16 (0.104) | 0.05 (0.105) | 0.00 (0.163)
  Weight deficit: Week 12 | 0.13 (0.066) | 0.20 (0.078) | 0.00 (0.100)
  Weight deficit: Week 24: number analyzed (Participants) | 12 | 18 | 15
  Weight deficit: Week 24 | 0.10 (0.102) | 0.29 (0.106) | 0.15 (0.124)
  BMI deficit: Week 12 | 0.18 (0.148) | 0.23 (0.114) | 0.08 (0.147)
  BMI deficit: Week 24: number analyzed (Participants) | 12 | 17 | 15
  BMI deficit: Week 24 | 0.26 (0.156) | 0.36 (0.113) | 0.20 (0.203)

6. Secondary Outcome: Percentage of Responders for Pruritus Assessments Based on Bi-Weekly and Monthly Scores Using the Albireo Observer-Reported Outcome Instrument at Weeks 12 and 24
Description: The responder for pruritus scores was defined as a participant who achieved at least a 1-point reduction in the ObsRO pruritus score. Percentages are rounded to hundredth decimal.
Time Frame: Weeks 12 and 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment. Only participants with data collected at specific timepoints are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
percentage of participants
  AM and PM scores combined: Week 12 (Bi-weekly score) | 5.0 [0.13 to 24.87] | 60.9 [38.54 to 80.29] | 42.1 [20.25 to 66.50]
  AM and PM scores combined: Week 12 (Monthly score) | 10.0 [1.23 to 31.70] | 52.2 [30.59 to 73.18] | 42.1 [20.25 to 66.50]
  AM and PM scores combined: Week 24 (Bi-weekly score): number analyzed (Participants) | 17 | 23 | 18
  AM and PM scores combined: Week 24 (Bi-weekly score) | 11.8 [1.46 to 36.44] | 43.5 [23.19 to 65.51] | 33.3 [13.34 to 59.01]
  AM and PM scores combined: Week 24 (Monthly score): number analyzed (Participants) | 19 | 23 | 19
  AM and PM scores combined: Week 24 (Monthly score) | 10.5 [1.30 to 33.14] | 52.2 [30.59 to 73.18] | 31.6 [12.58 to 56.55]
  AM score: Week 12 (Bi-weekly score) | 10.0 [1.23 to 31.70] | 60.9 [38.54 to 80.29] | 42.1 [20.25 to 66.50]
  AM score: Week 12 (Monthly score) | 10.0 [1.23 to 31.70] | 56.5 [34.49 to 76.81] | 42.1 [20.25 to 66.50]
  AM score: Week 24 (Bi-weekly score): number analyzed (Participants) | 17 | 23 | 18
  AM score: Week 24 (Bi-weekly score) | 11.8 [1.46 to 36.44] | 39.1 [19.71 to 61.46] | 33.3 [13.34 to 59.01]
  AM score: Week 24 (Monthly score): number analyzed (Participants) | 19 | 23 | 19
  AM score: Week 24 (Monthly score) | 15.8 [3.38 to 39.58] | 52.2 [30.59 to 73.18] | 42.1 [20.25 to 66.50]
  PM score: Week 12 (Bi-weekly score) | 10.0 [1.23 to 31.70] | 65.2 [42.73 to 83.62] | 36.8 [16.29 to 61.64]
  PM score: Week 12 (Monthly score) | 10.0 [1.23 to 31.70] | 60.9 [38.54 to 80.29] | 36.8 [16.29 to 61.64]
  PM score: Week 24 (Bi-weekly score): number analyzed (Participants) | 17 | 23 | 18
  PM score: Week 24 (Bi-weekly score) | 11.8 [1.46 to 36.44] | 56.5 [34.49 to 76.81] | 33.3 [13.34 to 59.01]
  PM score: Week 24 (Monthly score): number analyzed (Participants) | 19 | 23 | 19
  PM score: Week 24 (Monthly score) | 10.5 [1.30 to 33.14] | 52.2 [30.59 to 73.18] | 31.6 [12.58 to 56.55]

7. Secondary Outcome: Change From Baseline in Sleep Parameters Based on the Albireo Observer-reported Outcome Instrument Over the 24-Week Treatment Period
Description: The sleep disturbance were recorded twice daily via the electronic diary (eDiary). Participants and/or caregivers completed the eDiary every day in the morning and in the evening. The morning diary was completed shortly after the participant woke up and was used to record nighttime itching and scratching severity, aspects of sleep disturbance, and tiredness upon waking (AM scores). The evening/bedtime diary was completed just before the participant went to bed and recorded participant's itching and scratching severity, and tiredness during the day (PM scores). Both morning and bedtime diaries included Albireo ObsRO and PRO items. Baseline was the average of 14-day scores before the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 1 to 4, Weeks 5 to 8, Weeks 9 to 12, Weeks 13 to 16, Weeks 17 to 20, and Weeks 21 to 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
percentage of days
  Seeing blood due to scratching: Weeks 1 to 4 | -15.79 (4.700) | -14.42 (5.854) | -12.97 (6.036)
  Seeing blood due to scratching: Weeks 5 to 8: number analyzed (Participants) | 20 | 22 | 19
  Seeing blood due to scratching: Weeks 5 to 8 | -12.10 (6.353) | -26.22 (7.427) | -13.99 (7.770)
  Seeing blood due to scratching: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  Seeing blood due to scratching: Weeks 9 to 12 | -13.49 (6.320) | -29.22 (7.593) | -16.89 (9.258)
  Seeing blood due to scratching: Weeks 13 to 16: number analyzed (Participants) | 17 | 19 | 16
  Seeing blood due to scratching: Weeks 13 to 16 | -15.75 (6.264) | -33.38 (8.219) | -18.16 (9.403)
  Seeing blood due to scratching: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  Seeing blood due to scratching: Weeks 17 to 20 | -22.02 (7.999) | -32.14 (8.531) | -18.02 (9.967)
  Seeing blood due to scratching: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  Seeing blood due to scratching: Weeks 21 to 24 | -23.72 (8.563) | -30.82 (8.184) | -15.52 (10.465)
  Help falling asleep: Weeks 1 to 4 | -0.91 (1.596) | -14.73 (5.683) | -20.37 (6.390)
  Help falling asleep: Weeks 5 to 8: number analyzed (Participants) | 20 | 22 | 19
  Help falling asleep: Weeks 5 to 8 | -2.35 (2.397) | -25.03 (7.527) | -31.49 (10.209)
  Help falling asleep: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  Help falling asleep: Weeks 9 to 12 | -0.90 (1.152) | -31.03 (8.061) | -36.72 (11.154)
  Help falling asleep: Weeks 13 to 16: number analyzed (Participants) | 17 | 19 | 16
  Help falling asleep: Weeks 13 to 16 | -0.86 (1.392) | -46.10 (9.677) | -37.76 (12.013)
  Help falling asleep: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  Help falling asleep: Weeks 17 to 20 | -6.27 (3.862) | -45.65 (9.524) | -40.51 (12.566)
  Help falling asleep: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  Help falling asleep: Weeks 21 to 24 | -3.19 (2.890) | -51.75 (9.857) | -32.58 (14.573)
  Soothing: Weeks 1 to 4 | -1.15 (1.338) | -12.92 (5.911) | -21.88 (6.228)
  Soothing: Weeks 5 to 8: number analyzed (Participants) | 20 | 22 | 19
  Soothing: Weeks 5 to 8 | -3.76 (2.773) | -17.89 (7.562) | -35.97 (9.795)
  Soothing: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  Soothing: Weeks 9 to 12 | -5.00 (2.819) | -29.79 (8.570) | -41.21 (10.796)
  Soothing: Weeks 13 to 16: number analyzed (Participants) | 17 | 19 | 16
  Soothing: Weeks 13 to 16 | -2.12 (3.006) | -42.79 (10.364) | -40.23 (11.611)
  Soothing: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  Soothing: Weeks 17 to 20 | -4.73 (3.742) | -44.96 (10.485) | -40.13 (12.324)
  Soothing: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  Soothing: Weeks 21 to 24 | -7.64 (6.182) | -51.48 (10.323) | -34.87 (13.369)
  Sleeping with the caregiver: Weeks 1 to 4 | -4.49 (1.961) | -15.30 (6.396) | -24.57 (7.024)
  Sleeping with the caregiver: Weeks 5 to 8: number analyzed (Participants) | 20 | 22 | 19
  Sleeping with the caregiver: Weeks 5 to 8 | -5.93 (3.649) | -19.73 (7.061) | -35.58 (10.053)
  Sleeping with the caregiver: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  Sleeping with the caregiver: Weeks 9 to 12 | -5.74 (3.585) | -26.12 (9.543) | -36.00 (10.361)
  Sleeping with the caregiver: Weeks 13 to 16: number analyzed (Participants) | 17 | 19 | 16
  Sleeping with the caregiver: Weeks 13 to 16 | -4.96 (3.481) | -40.55 (10.501) | -37.52 (11.083)
  Sleeping with the caregiver: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  Sleeping with the caregiver: Weeks 17 to 20 | -2.59 (3.688) | -42.20 (10.247) | -35.14 (11.563)
  Sleeping with the caregiver: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  Sleeping with the caregiver: Weeks 21 to 24 | -5.45 (4.844) | -49.35 (10.466) | -33.14 (11.801)
  Taking medications to induce sleep: Weeks 1 to 4 | -1.78 (1.921) | -0.61 (1.913) | 0.98 (2.320)
  Taking medications to induce sleep: Weeks 5 to 8: number analyzed (Participants) | 20 | 22 | 19
  Taking medications to induce sleep: Weeks 5 to 8 | 1.44 (4.292) | 0.18 (3.018) | -2.43 (3.036)
  Taking medications to induce sleep: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  Taking medications to induce sleep: Weeks 9 to 12 | 2.40 (4.271) | 1.31 (3.656) | -5.74 (4.967)
  Taking medications to induce sleep: Weeks 13 to 16: number analyzed (Participants) | 17 | 19 | 16
  Taking medications to induce sleep: Weeks 13 to 16 | 0.16 (4.647) | -1.61 (2.556) | -4.58 (4.681)
  Taking medications to induce sleep: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  Taking medications to induce sleep: Weeks 17 to 20 | 3.53 (5.384) | -1.99 (2.141) | -3.26 (6.403)
  Taking medications to induce sleep: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  Taking medications to induce sleep: Weeks 21 to 24 | 5.50 (5.307) | -0.03 (2.251) | 2.04 (8.413)

8. Secondary Outcome: Change From Baseline in Sleep Parameters Based on the Albireo Patient-Reported Outcome (PRO) Instrument Over the 24-Week Treatment Period
Description: The ObsRO and electronic diary (eDiary) PRO scale called PRUCISION was used to assess pruritus and sleep outcomes. Participants and/or caregivers completed the eDiary every day in the morning (AM scores) and in the evening (PM scores). Specifically, for difficulty falling or staying asleep, the following 2 respective questions were asked in the Morning Daily eDiary: 1) How hard was it to fall asleep last night because of your itching. and 2) How hard was it to stay asleep last night because of your itching. The PRO was a 5-point scale, and scores ranged from 0 (no itching) to 28 (the worst itching), where higher scores indicated a greater amount of itching, sleep disturbance, and tiredness. No subscales were used. Change in sleep parameters measured with the Albireo PRO and ObsRO instruments by each 4-week interval over the 24-week treatment period was assessed. Baseline was the average of 14-day scores before the first dose of study treatment.
Time Frame: Baseline (Day 1) and Weeks 1 to 4, Weeks 5 to 8, Weeks 9 to 12, Weeks 13 to 16, Weeks 17 to 20, and Weeks 21 to 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 2 | 2 | 5
scores on a scale
  Difficulty falling asleep: Weeks 1 to 4 | -0.46 (0.143) | -0.72 (0.494) | -0.59 (0.394)
  Difficulty falling asleep: Weeks 5 to 8 | -0.34 (0.018) | -1.40 (1.009) | -0.65 (0.571)
  Difficulty falling asleep: Weeks 9 to 12 | -0.38 (0.339) | -2.31 (0.499) | -0.95 (0.650)
  Difficulty falling asleep: Weeks 13 to 16 | -0.16 (0.268) | -2.07 (0.863) | -1.01 (0.665)
  Difficulty falling asleep: Weeks 17 to 20 | -0.52 (0.228) | -2.12 (0.974) | -1.02 (0.710)
  Difficulty falling asleep: Weeks 21 to 24 | -0.25 (0.179) | -2.22 (0.823) | -0.82 (0.658)
  Difficulty staying asleep: Weeks 1 to 4 | -0.13 (0.411) | -0.70 (0.548) | -0.43 (0.440)
  Difficulty staying asleep: Weeks 5 to 8 | 0.09 (0.518) | -1.48 (0.932) | -0.50 (0.553)
  Difficulty staying asleep: Weeks 9 to 12 | 0.02 (0.661) | -2.51 (0.352) | -0.77 (0.670)
  Difficulty staying asleep: Weeks 13 to 16 | 0.13 (0.625) | -2.46 (0.464) | -0.89 (0.626)
  Difficulty staying asleep: Weeks 17 to 20 | -0.15 (0.147) | -2.36 (0.637) | -0.95 (0.644)
  Difficulty staying asleep: Weeks 21 to 24 | 0.25 (0.429) | -2.55 (0.448) | -0.78 (0.633)

9. Secondary Outcome: Percentage of Individual Assessments Meeting the Definition of a Positive Pruritus Assessment at the Participant Level Using the Albireo ObsRO Instrument Over the 24-Week Treatment Period
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least 1 point drop from baseline based on the Albireo ObsRO instrument. The percentage of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant multiplied by 100. At each assessment, the AM or PM score was compared to the baseline AM or PM average, respectively.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Error); unit: percentage of assessments
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
percentage of assessments
  AM and PM scores combined: Weeks 0 to 4 | 33.48 (5.881) | 51.40 (5.818) | 42.48 (7.508)
  AM and PM scores combined: Weeks 0 to 8 | 32.72 (5.871) | 54.23 (5.887) | 48.21 (7.479)
  AM and PM scores combined: Weeks 0 to 12 | 32.35 (5.945) | 58.85 (5.738) | 49.15 (7.428)
  AM and PM scores combined: Weeks 0 to 16 | 30.67 (5.522) | 58.83 (5.925) | 48.31 (7.624)
  AM and PM scores combined: Weeks 0 to 18 | 29.88 (5.462) | 58.80 (6.004) | 48.25 (7.809)
  AM and PM scores combined: Weeks 0 to 20 | 29.45 (5.376) | 58.68 (6.079) | 48.10 (7.975)
  AM score: Weeks 0 to 4 | 31.07 (5.436) | 48.14 (6.161) | 47.37 (8.439)
  AM score: Weeks 0 to 8 | 31.07 (5.213) | 51.16 (6.129) | 51.79 (8.001)
  AM score: Weeks 0 to 12 | 31.07 (5.374) | 56.06 (5.922) | 52.26 (7.693)
  AM score: Weeks 0 to 16 | 29.91 (5.246) | 56.41 (6.183) | 50.47 (7.660)
  AM score: Weeks 0 to 18 | 28.93 (5.224) | 56.35 (6.249) | 49.92 (7.800)
  AM score: Weeks 0 to 20 | 28.50 (5.206) | 56.27 (6.293) | 49.74 (7.993)
  AM score: Weeks 0 to 24 | 28.17 (5.276) | 55.73 (6.396) | 48.92 (8.197)
  PM score: Weeks 0 to 4 | 35.89 (7.055) | 54.66 (6.594) | 37.59 (7.629)
  PM score: Weeks 0 to 8 | 34.38 (7.290) | 57.30 (6.478) | 44.64 (7.804)
  PM score: Weeks 0 to 12 | 33.63 (7.404) | 61.65 (6.330) | 46.05 (7.884)
  PM score: Weeks 0 to 16 | 31.43 (7.006) | 61.26 (6.205) | 46.15 (8.178)
  PM score: Weeks 0 to 18 | 30.83 (6.898) | 61.25 (6.225) | 46.57 (8.363)
  PM score: Weeks 0 to 20 | 30.39 (6.812) | 61.09 (6.284) | 46.47 (8.434)
  PM score: Weeks 0 to 24 | 29.31 (6.592) | 60.89 (6.385) | 46.47 (8.456)

10. Secondary Outcome: Percentage of Individual Assessments Meeting the Definition of a Positive Pruritus Assessment at the Participant Level Using the Albireo PRO Instrument Over the 24-Week Treatment Period
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least 1 point drop from baseline based on the Albireo PRO instrument, only participants >=8 years of age completed the Albireo PRO instrument. The percentage of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant multiplied by 100. At each assessment, the AM or PM score was compared to the baseline AM or PM average, respectively.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Mean (Standard Error); unit: percentage of assessments
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 2 | 2 | 5
percentage of assessments
  AM and PM scores combined: Weeks 0 to 4 | 64.29 (8.929) | 43.75 (25.893) | 38.93 (15.272)
  AM and PM scores combined: Weeks 0 to 8 | 46.88 (12.946) | 52.68 (25.893) | 41.96 (16.178)
  AM and PM scores combined: Weeks 0 to 12 | 41.96 (10.417) | 63.39 (18.155) | 45.00 (16.939)
  AM and PM scores combined: Weeks 0 to 16 | 38.62 (3.348) | 66.74 (18.080) | 46.96 (17.477)
  AM and PM scores combined: Weeks 0 to 18 | 37.50 (0.198) | 67.66 (18.849) | 47.14 (17.558)
  AM and PM scores combined: Weeks 0 to 20 | 34.82 (0.179) | 67.32 (20.179) | 48.07 (18.010)
  AM and PM scores combined: Weeks 0 to 24 | 31.70 (1.637) | 68.88 (19.772) | 47.65 (17.997)
  AM score: Weeks 0 to 4 | 55.36 (8.929) | 41.07 (23.214) | 37.86 (16.115)
  AM score: Weeks 0 to 8 | 39.29 (14.286) | 50.00 (21.429) | 38.93 (16.243)
  AM score: Weeks 0 to 12 | 33.93 (10.119) | 61.31 (11.310) | 41.43 (16.562)
  AM score: Weeks 0 to 16 | 31.70 (1.339) | 65.18 (12.500) | 42.68 (16.554)
  AM score: Weeks 0 to 18 | 31.35 (1.190) | 66.67 (13.492) | 42.22 (16.343)
  AM score: Weeks 0 to 20 | 28.93 (0.357) | 66.07 (15.357) | 43.71 (16.860)
  AM score: Weeks 0 to 24 | 26.19 (1.190) | 66.72 (16.718) | 43.24 (16.835)
  PM score: Weeks 0 to 4 | 73.21 (8.929) | 46.43 (28.571) | 40.00 (15.042)
  PM score: Weeks 0 to 8 | 54.46 (11.607) | 55.36 (30.357) | 45.00 (16.545)
  PM score: Weeks 0 to 12 | 50.00 (10.714) | 65.48 (25.000) | 48.57 (17.715)
  PM score: Weeks 0 to 16 | 45.54 (5.357) | 68.30 (23.661) | 51.25 (18.751)
  PM score: Weeks 0 to 18 | 43.65 (1.587) | 68.65 (24.206) | 52.06 (19.230)
  PM score: Weeks 0 to 20 | 40.71 (0.000) | 68.57 (25.000) | 52.43 (19.568)
  PM score: Weeks 0 to 24 | 37.20 (2.083) | 71.04 (22.825) | 52.06 (19.595)

11. Secondary Outcome: Percentage of Individual Assessments Meeting the Definition of a Positive Pruritus Assessment at the Participant Level Using the Albireo ObsRO Instrument Over the 24-Week Treatment Period
Description: as for outcome 9
Time Frame: Baseline (Day 1) and Weeks 1 to 4, Weeks 5 to 8, Weeks 9 to 12, Weeks 13 to 16, Weeks 17 to 20, and Weeks 21 to 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: percentage of assessments
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
percentage of assessments
  AM and PM scores combined: Weeks 1 to 4 | 33.48 (5.881) | 51.40 (5.818) | 42.48 (7.508)
  AM and PM scores combined: Weeks 5 to 8 | 31.96 (6.515) | 57.07 (6.714) | 53.95 (8.423)
  AM and PM scores combined: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  AM and PM scores combined: Weeks 9 to 12 | 31.61 (6.794) | 68.09 (6.357) | 53.67 (9.404)
  AM and PM scores combined: Weeks 13 to 16: number analyzed (Participants) | 17 | 20 | 16
  AM and PM scores combined: Weeks 13 to 16 | 28.36 (7.534) | 67.59 (7.779) | 54.35 (9.802)
  AM and PM scores combined: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  AM and PM scores combined: Weeks 17 to 20 | 32.62 (8.583) | 66.79 (7.805) | 56.14 (10.655)
  AM and PM scores combined: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  AM and PM scores combined: Weeks 21 to 24 | 35.42 (8.783) | 68.57 (6.926) | 55.12 (10.047)
  AM score: Weeks 1 to 4 | 31.07 (5.436) | 48.14 (6.161) | 47.37 (8.439)
  AM score: Weeks 5 to 8 | 31.07 (5.812) | 54.19 (6.783) | 56.20 (8.483)
  AM score: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  AM score: Weeks 9 to 12 | 31.07 (6.747) | 65.84 (6.854) | 55.95 (9.383)
  AM score: Weeks 13 to 16: number analyzed (Participants) | 17 | 20 | 16
  AM score: Weeks 13 to 16 | 29.62 (8.502) | 66.07 (8.042) | 53.57 (9.550)
  AM score: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  AM score: Weeks 17 to 20 | 30.24 (8.733) | 64.11 (8.121) | 55.58 (11.171)
  AM score: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  AM score: Weeks 21 to 24 | 37.30 (10.909) | 64.37 (7.324) | 54.35 (10.801)
  PM score: Weeks 1 to 4 | 35.89 (7.055) | 54.66 (6.594) | 37.59 (7.629)
  PM score: Weeks 5 to 8 | 32.86 (8.138) | 59.94 (7.355) | 51.69 (9.051)
  PM score: Weeks 9 to 12: number analyzed (Participants) | 20 | 23 | 18
  PM score: Weeks 9 to 12 | 32.14 (8.078) | 70.34 (6.816) | 51.39 (10.015)
  PM score: Weeks 13 to 16: number analyzed (Participants) | 17 | 20 | 16
  PM score: Weeks 13 to 16 | 27.10 (8.997) | 69.11 (7.783) | 55.13 (10.664)
  PM score: Weeks 17 to 20: number analyzed (Participants) | 15 | 20 | 16
  PM score: Weeks 17 to 20 | 35.00 (10.323) | 69.46 (7.848) | 56.70 (10.554)
  PM score: Weeks 21 to 24: number analyzed (Participants) | 14 | 19 | 16
  PM score: Weeks 21 to 24 | 33.54 (9.699) | 72.76 (7.185) | 55.90 (9.976)

12. Secondary Outcome: Number of Participants Underwent Biliary Diversion Surgery and Liver Transplantation
Description: The number of participants underwent biliary diversion surgery and liver transplantation was determined.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
Participants
  Biliary diversion surgery | 0 | 0 | 0
  Liver transplantation | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Achieved Positive Pruritus Assessment for >50% of the Time Based on the Albireo ObsRO and PRO Instruments Over the 24-Week Treatment Period
Description: A positive pruritus assessment was defined as a scratching score of <=1 or at least 1 point drop from baseline based on the Albireo ObsRO and PRO instruments. The percentage of positive pruritus assessment was calculated as the number of positive pruritus assessments divided by the total number of reported assessments only when more than 50% of planned assessment recorded by each participant multiplied by 100.
Time Frame: From Baseline (Day 1) up to Week 24
Population: The FAS included all randomized participants who received at least 1 dose of study treatment. Only participants with data collected for specific instrument are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
Number analyzed (Participants) | 20 | 23 | 19
Participants
  Albireo ObsRO Instrument: AM and PM scores combined | 4 | 17 | 9
  Albireo ObsRO Instrument: AM score | 3 | 13 | 10
  Albireo ObsRO Instrument: PM score | 5 | 16 | 9
  Albireo PRO Instrument: AM and PM scores combined: number analyzed (Participants) | 2 | 2 | 5
  Albireo PRO Instrument: AM and PM scores combined | 0 | 1 | 3
  Albireo PRO Instrument: AM score: number analyzed (Participants) | 2 | 2 | 5
  Albireo PRO Instrument: AM score | 0 | 1 | 3
  Albireo PRO Instrument: PM score: number analyzed (Participants) | 2 | 2 | 5
  Albireo PRO Instrument: PM score | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: All serious and non-serious adverse events (AEs) were collected once the caregiver/participant had signed the informed consent form (ICF) and until the post-treatment follow-up (Visit 10) or 28 days after the last dose of study treatment, approximately 28 weeks
Description: Treatment emergent adverse events were defined as any AE that occurred after first dose or AE occurred before first dose but worsened in severity on or after first dose. Treatment emergent serious adverse events and treatment emergent non-serious AEs are reported here.
Arm/Group | Placebo | A4250 Low Dose | A4250 High Dose
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/23 | 0/19
Serious Adverse Events (participants affected / at risk) | 5/20 | 0/23 | 3/19
Other Adverse Events (participants affected / at risk) | 17/20 | 19/23 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | A4250 Low Dose (N=23) | A4250 High Dose (N=19)
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Gastroenteritis adenovirus (Infections and infestations) | 1 | 0 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Auricular haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Weight gain poor (Metabolism and nutrition disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=20) | A4250 Low Dose (N=23) | A4250 High Dose (N=19)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 9 | 4
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 4 | 3
Influenza like illness (General disorders) | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 5 | 7 | 5
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2
Otitis media (Infections and infestations) | 0 | 0 | 2
Parotitis (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Viral diarrhoea (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1
Viral rash (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Auricular haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 2 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 1
Bilirubin conjugated increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 2
Blood bilirubin increased (Investigations) | 2 | 3 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 1
Blood creatinine decreased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0
Liver palpable (Investigations) | 0 | 1 | 0
Platelet count increased (Investigations) | 1 | 0 | 1
Product residue present (Investigations) | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1
Vitamin E increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin A deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 2
Vitamin E deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Irritability (Psychiatric disorders) | 1 | 0 | 1
Selective eating disorder (Psychiatric disorders) | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 1
Skin candida (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Albireo will retain the ownership of all data. All proposed publications based on this study must be subject to the sponsor's approval requirements.

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03566238/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT03566238/SAP_001.pdf